CLINICAL TRIAL: NCT04674254
Title: Macular Perfusion Changes in Proliferative Diabetic Retinopathy Following Anti-VEGF Therapy Versus Targeted and Pan-retinal Photocoagulation Using Optical Coherence Tomography Angiography
Brief Title: Macular Perfusion Changes After Anti-VEGF Versus Targeted Retinal Photocoagulation in Proliferative Diabetic Retinopathy
Acronym: PROPER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ayman Gehad Elnahry, Lecturer of Ophthalmology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MD-39-2021
Record Dates: First submitted 2020-12-06; First posted 2020-12-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Proliferative Diabetic Retinopathy; Vascular Endothelial Growth Factor Overexpression; Diabetic Retinopathy
Keywords: Proliferative diabetic retinopathy; anti-vascular endothelial growth factor; optical coherence tomography angiography; macular perfusion; pan-retinal photocoagulation; fluorescein angiography; visual field
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Anti-vascular endothelial growth factor agent (Active Comparator): Intravitreal injections of 1.25 mg/0.05 ml of Bevacizumab every 4 weeks through 12- week visit then pro re nata to complete 12 months according to Protocol S.
  Interventions: Drug: Bevacizumab Injection
- Targeted retinal photocoagulation (Active Comparator): Targeted retinal photocoagulation guided by fundus fluorescein angiography will be administered after topical anesthesia, directed to areas of nonperfused peripheral retina plus a 1-disc area margin using the Mainster lens. Subsequent treatments if needed will be delivered at 3 monthly intervals for a minimum follow-up of 12 months. The extent of the laser applied will be determined based on areas of nonperfusion identified by fundus fluorescein angiography.
  Interventions: Procedure: Targeted retinal photocoagulation
- Standard pan-retinal photocoagulation (Active Comparator): Standard pan-retinal photocoagulation will be performed at baseline and then every 3 months thereafter if needed, for a minimum follow-up period of 12 months.
  PRP will be performed at two consecutive sessions with adherence to the guidelines of the Early Treatment Diabetic Retinopathy Study Group. Following topical anesthesia, 1000 to 1200 laser spots will be applied to the retina at each session with a 532 nm frequency doubled Nd-YAG laser (VISULAS, Carl Zeiss, Germany) using a spot size of 300-500 μm. PRP will be applied in all 4 retina quadrants.
  The Mainster lens will be used. Retreatment will be done according to the Diabetic Retinopathy Clinical Research network protocol S classification for patients with stable, worsening, or with failure of regression of neovascularization.
  Interventions: Procedure: Standard pan-retinal photocoagulation

INTERVENTIONS:
Drug: Bevacizumab Injection — Bevacizumab will be intravitreally injected every 4 weeks through 12 weeks then pro re nata thereafter for 12 months.
  Other Names: Avastin
  Arms: Anti-vascular endothelial growth factor agent
Procedure: Targeted retinal photocoagulation — Targeted retinal photocoagulation will be administered to nonperfused areas detected on fundus fluorescein angiography at baseline and repeated every 3 months as needed for 12 months.
  Arms: Targeted retinal photocoagulation
Procedure: Standard pan-retinal photocoagulation — Standard pan-retinal photocoagulation will be applied to perfused and nonperfused areas of the retinal periphery at baseline and every 3 months as needed for 12 months.
  Arms: Standard pan-retinal photocoagulation

SUMMARY:
Diabetic retinopathy (DR) is the most common microvascular complication of diabetes mellitus (DM), while proliferative diabetic retinopathy (PDR) is the principal cause of severe visual loss in patients with diabetes. Since 1981, Panretinal photocoagulation (PRP) has been a standard of treatment for PDR. However, PRP can be associated with adverse effects, including visual field constriction, decreased night vision, and worsening of coexisting diabetic macular edema (DME). For this reason, some authors have advocated targeted treatment with PRP. Targeted retinal laser photocoagulation (TRP) is designed to treat areas of retinal capillary non-perfusion and intermediate retinal ischemic zones in PDR that may spare better-perfused tissue from laser-induced tissue scarring.

Protocol S by Diabetic Retinopathy Clinical Research Network (DRCR.net) has shown that patients that receive ranibizumab as anti-vascular endothelial growth factor (anti-VEGF) therapy with deferred PRP are non-inferior regarding improving in visual acuity to those eyes receiving standard prompt PRP therapy for the treatment of PDR.

Retinal ischemia is an important factor in the progression and prognosis of diabetic retinopathy. Regarding the effect of anti-VEGF drugs on macular perfusion, several studies have shown mixed results with an increase, decrease, or no effect on perfusion in response to anti-VEGF treatment. In many of these studies, however, patients with more ischemic retinas were not included. Fluorescein angiography (FA) was the method used to assess changes in macular perfusion after anti-VEGF injections in most of the clinical trials. Despite its clinical usefulness, however, FA is known to have documented risks. Optical coherence tomography angiography (OCTA) in macular perfusion evaluation in these cases was recommended by some investigators. Several studies have proved the reliability of OCTA in detecting and quantifying macular ischemia in diabetics.

The investigators aim to compare changes in the macular perfusion in patients with PDR after treatment with anti-VEGF therapy versus TRP versus Standard PRP using OCTA.

DETAILED DESCRIPTION:
Diabetic retinopathy (DR) is the most common microvascular complication of diabetes mellitus (DM), while proliferative diabetic retinopathy (PDR) is the principal cause of severe visual loss in patients with diabetes.

Since 1981, PRP has been a standard of treatment for PDR. However, PRP can be associated with adverse effects, including visual field constriction, decreased night vision, and worsening of coexisting diabetic macular edema (DME). for this reason, some authors have advocated targeted treatment with PRP. Targeted retinal laser photocoagulation (TRP) is designed to treat areas of retinal capillary non-perfusion and intermediate retinal ischemic zones in PDR that may spare better-perfused tissue from laser-induced tissue scarring.

Protocol S by DRCR.net has shown that patients that receive ranibizumab as anti-vascular endothelial growth factor (anti-VEGF) therapy with deferred PRP are non-inferior regarding improving in visual acuity to those eyes receiving standard prompt PRP therapy for the treatment of PDR. However, the effect of both treatment modalities on macular perfusion has been inconclusive with no studies comparing the effect of both.

Regarding the effect of anti-VEGF drugs on macular perfusion, several studies have shown mixed results with an increase, decrease, or no effect on perfusion in response to anti-VEGF treatment. In many of these studies, however, patients with more ischemic retinas were not included. Retinal ischemia is an important factor in the progression and prognosis of diabetic retinopathy.

Fluorescein angiography (FA) was the method used to assess changes in macular perfusion after anti-VEGF injections in most of the clinical trials. Despite its clinical usefulness, however, FA is known to have documented risks and is being replaced by optical coherence tomography angiography (OCTA) in macular perfusion evaluation in these cases.

OCTA is a new noninvasive method of acquiring high-resolution images of the retinal vasculature that can be utilized in the management and study of retinal diseases without the need for dye injection. It allows the visualization of both the superficial and deep retinal capillary layers separately and the construction of microvascular flow maps allowing quantitative analysis of vascular parameters.

OCTA uses high-speed OCT scanning to detect the flow of blood by analyzing signal decorrelation between two sequential OCT cross-sectional scans repeated at the same location. Because of the movement of erythrocytes within a vessel, compared to stationary areas of the surrounding retina, only perfused blood vessels will result in signal decorrelation, leading to their imaging. The split-spectrum amplitude-decorrelation angiography (SSADA) algorithm improves the signal to noise ratio.

Several studies have proved the reliability of OCTA in detecting and quantifying macular ischemia in diabetics.

The investigators aim to compare changes in the macular perfusion in patients with PDR without macular edema after treatment with anti-VEGF therapy versus TRP versus Standard PRP using OCTA.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years old
2. Type 1 or 2 diabetes mellitus
3. PDR
4. Central macular thickness less than 300 µm

Exclusion Criteria:

1. Central macular thickness more than 300 µm
2. Previous retinal laser treatment
3. Ocular conditions that may affect macular perfusion (e.g. retinal vein occlusion, uveitis, vasculitis etc.)
4. Any previous treatment for diabetic macular edema.
5. Presence of epiretinal membrane involving the macula or vitreomacular traction
6. Media opacity such vitreous hemorrhage and dense cataract.
7. Patients with previous cataract surgery within the last 3 months.
8. Uncontrolled glaucoma
9. Thromboembolic events within 6 months
10. Tractional retinal detachment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Change in foveal avascular zone area | 0, 3, 6, 9, and 12 months
  The change in the foveal avascular zone area will be compared between the different treatment arms as a measure of macular perfusion change.
Change in vascular density of the retinal capillary plexuses | 0, 3, 6, 9, and 12 months
  The change in retinal capillary vascular densities at different capillary layers will be compared between the different treatment arms as a measure of macular perfusion change.

SECONDARY OUTCOMES:
Change in neovessels | 0, 3, 6, 9, and 12 months
  The change in neovessels following treatment with each modality will be evaluated clinically and by fundus fluorescein angiography and the response to treatment will be classified according to the criteria of protocol S of the DRCR network
Change in central macular thickness | 0, 3, 6, 9, and 12 months
  The change in central macular thickness will be evaluated following treatment with each modality using optical coherence tomography.
Change in best corrected visual acuity | 0, 3, 6, 9, and 12 months
  The change in best corrected visual acuity will be assessed following treatment with each modality using standard Snellen charts.
Change in macular sensitivity | 0, 3, 6, 9, and 12 months
  The change in the macular sensitivity will be assessed following treatment with each modality using macular microperimetry.
Change in orbital blood flow | 0, 3, 6, 9, and 12 months
  The change in orbital blood flow will be assessed following treatment with each modality using orbital color duplex imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Eldaly, MD, PhD, Study Chair — Cairo University; Ayman G Elnahry, MD, PhD, Principal Investigator — Cairo University; Wael A Yussuf, MD, MSc, Study Director — Cairo University; Ahmed A Abdel-Kader, MD, PhD, Study Director — Cairo University; Ahmed A Mohalhal, MD, PhD, Study Director — Cairo University
Locations (1):
- Faculty of Medicine, Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No
Results will be posted on clinicaltrials.gov when the study is concluded.

REFERENCES:
- [Result] Lee R, Wong TY, Sabanayagam C. Epidemiology of diabetic retinopathy, diabetic macular edema and related vision loss. Eye Vis (Lond). 2015 Sep 30;2:17. doi: 10.1186/s40662-015-0026-2. eCollection 2015. PMID 26605370
- [Result] Klein R, Klein BE, Moss SE, Davis MD, DeMets DL. The Wisconsin epidemiologic study of diabetic retinopathy. IV. Diabetic macular edema. Ophthalmology. 1984 Dec;91(12):1464-74. doi: 10.1016/s0161-6420(84)34102-1. PMID 6521986
- [Result] Riaskoff S. Photocoagulation treatment of proliferative diabetic retinopathy. Bull Soc Belge Ophtalmol. 1981;197:9-17. No abstract available. PMID 6182936
- [Result] Alagorie AR, Nittala MG, Velaga S, Zhou B, Rusakevich AM, Wykoff CC, Sadda SR. Association of Intravitreal Aflibercept With Optical Coherence Tomography Angiography Vessel Density in Patients With Proliferative Diabetic Retinopathy: A Secondary Analysis of a Randomized Clinical Trial. JAMA Ophthalmol. 2020 Aug 1;138(8):851-857. doi: 10.1001/jamaophthalmol.2020.2130. PMID 32584384
- [Result] Muqit MM, Marcellino GR, Henson DB, Young LB, Patton N, Charles SJ, Turner GS, Stanga PE. Optos-guided pattern scan laser (Pascal)-targeted retinal photocoagulation in proliferative diabetic retinopathy. Acta Ophthalmol. 2013 May;91(3):251-8. doi: 10.1111/j.1755-3768.2011.02307.x. Epub 2011 Dec 16. PMID 22176513
- [Result] Nikkhah H, Ghazi H, Razzaghi MR, Karimi S, Ramezani A, Soheilian M. Extended targeted retinal photocoagulation versus conventional pan-retinal photocoagulation for proliferative diabetic retinopathy in a randomized clinical trial. Int Ophthalmol. 2018 Feb;38(1):313-321. doi: 10.1007/s10792-017-0469-7. Epub 2017 Feb 6. PMID 28168567
- [Result] Wessel MM, Aaker GD, Parlitsis G, Cho M, D'Amico DJ, Kiss S. Ultra-wide-field angiography improves the detection and classification of diabetic retinopathy. Retina. 2012 Apr;32(4):785-91. doi: 10.1097/IAE.0b013e3182278b64. PMID 22080911
- [Result] Kozak I, Luttrull JK. Modern retinal laser therapy. Saudi J Ophthalmol. 2015 Apr-Jun;29(2):137-46. doi: 10.1016/j.sjopt.2014.09.001. Epub 2014 Sep 28. PMID 25892934
- [Result] Writing Committee for the Diabetic Retinopathy Clinical Research Network; Gross JG, Glassman AR, Jampol LM, Inusah S, Aiello LP, Antoszyk AN, Baker CW, Berger BB, Bressler NM, Browning D, Elman MJ, Ferris FL 3rd, Friedman SM, Marcus DM, Melia M, Stockdale CR, Sun JK, Beck RW. Panretinal Photocoagulation vs Intravitreous Ranibizumab for Proliferative Diabetic Retinopathy: A Randomized Clinical Trial. JAMA. 2015 Nov 24;314(20):2137-2146. doi: 10.1001/jama.2015.15217. PMID 26565927
- [Result] Elnahry AG, Abdel-Kader AA, Raafat KA, Elrakhawy K. Evaluation of Changes in Macular Perfusion Detected by Optical Coherence Tomography Angiography following 3 Intravitreal Monthly Bevacizumab Injections for Diabetic Macular Edema in the IMPACT Study. J Ophthalmol. 2020 Apr 27;2020:5814165. doi: 10.1155/2020/5814165. eCollection 2020. PMID 32411431
- [Result] Elnahry AG, Abdel-Kader AA, Habib AE, Elnahry GA, Raafat KA, Elrakhawy K. Review on Recent Trials Evaluating the Effect of Intravitreal Injections of Anti-VEGF Agents on the Macular Perfusion of Diabetic Patients with Diabetic Macular Edema. Rev Recent Clin Trials. 2020;15(3):188-198. doi: 10.2174/1574887115666200519073704. PMID 32427087
- [Result] Elnahry AG, Abdel-Kader AA, Raafat KA, Elrakhawy K. Evaluation of the Effect of Repeated Intravitreal Bevacizumab Injections on the Macular Microvasculature of a Diabetic Patient Using Optical Coherence Tomography Angiography. Case Rep Ophthalmol Med. 2019 Apr 18;2019:3936168. doi: 10.1155/2019/3936168. eCollection 2019. PMID 31139483
- [Result] Ghasemi Falavarjani K, Iafe NA, Hubschman JP, Tsui I, Sadda SR, Sarraf D. Optical Coherence Tomography Angiography Analysis of the Foveal Avascular Zone and Macular Vessel Density After Anti-VEGF Therapy in Eyes With Diabetic Macular Edema and Retinal Vein Occlusion. Invest Ophthalmol Vis Sci. 2017 Jan 1;58(1):30-34. doi: 10.1167/iovs.16-20579. PMID 28114569
- [Result] Manousaridis K, Talks J. Macular ischaemia: a contraindication for anti-VEGF treatment in retinal vascular disease? Br J Ophthalmol. 2012 Feb;96(2):179-84. doi: 10.1136/bjophthalmol-2011-301087. PMID 22250209
- [Result] Hsieh YT, Alam MN, Le D, Hsiao CC, Yang CH, Chao DL, Yao X. OCT Angiography Biomarkers for Predicting Visual Outcomes after Ranibizumab Treatment for Diabetic Macular Edema. Ophthalmol Retina. 2019 Oct;3(10):826-834. doi: 10.1016/j.oret.2019.04.027. Epub 2019 May 7. PMID 31227330
- [Result] Michaelides M, Kaines A, Hamilton RD, Fraser-Bell S, Rajendram R, Quhill F, Boos CJ, Xing W, Egan C, Peto T, Bunce C, Leslie RD, Hykin PG. A prospective randomized trial of intravitreal bevacizumab or laser therapy in the management of diabetic macular edema (BOLT study) 12-month data: report 2. Ophthalmology. 2010 Jun;117(6):1078-1086.e2. doi: 10.1016/j.ophtha.2010.03.045. Epub 2010 Apr 22. PMID 20416952
- [Result] Nguyen QD, Brown DM, Marcus DM, Boyer DS, Patel S, Feiner L, Gibson A, Sy J, Rundle AC, Hopkins JJ, Rubio RG, Ehrlich JS; RISE and RIDE Research Group. Ranibizumab for diabetic macular edema: results from 2 phase III randomized trials: RISE and RIDE. Ophthalmology. 2012 Apr;119(4):789-801. doi: 10.1016/j.ophtha.2011.12.039. Epub 2012 Feb 11. PMID 22330964
- [Result] Campochiaro PA, Wykoff CC, Shapiro H, Rubio RG, Ehrlich JS. Neutralization of vascular endothelial growth factor slows progression of retinal nonperfusion in patients with diabetic macular edema. Ophthalmology. 2014 Sep;121(9):1783-9. doi: 10.1016/j.ophtha.2014.03.021. Epub 2014 Apr 24. PMID 24768239
- [Result] Yannuzzi LA, Rohrer KT, Tindel LJ, Sobel RS, Costanza MA, Shields W, Zang E. Fluorescein angiography complication survey. Ophthalmology. 1986 May;93(5):611-7. doi: 10.1016/s0161-6420(86)33697-2. PMID 3523356
- [Result] Freiberg FJ, Pfau M, Wons J, Wirth MA, Becker MD, Michels S. Optical coherence tomography angiography of the foveal avascular zone in diabetic retinopathy. Graefes Arch Clin Exp Ophthalmol. 2016 Jun;254(6):1051-8. doi: 10.1007/s00417-015-3148-2. Epub 2015 Sep 4. PMID 26338819
- [Result] Bradley PD, Sim DA, Keane PA, Cardoso J, Agrawal R, Tufail A, Egan CA. The Evaluation of Diabetic Macular Ischemia Using Optical Coherence Tomography Angiography. Invest Ophthalmol Vis Sci. 2016 Feb;57(2):626-31. doi: 10.1167/iovs.15-18034. PMID 26903223